

# STATISTICAL ANALYSIS PLAN

Title An Open-Label, Single-Arm, Phase 3 Study to Evaluate

the Effects of KRN23 on Osteomalacia in Adults with X-

linked Hypophosphatemia (XLH)

**Protocol:** UX023-CL304

Investigational Product: KRN23 (Recombinant human IgG1 monoclonal antibody

to fibroblast growth factor 23 [FGF23])

**Indication:** X-linked Hypophosphatemia (XLH)

**IND Number:** 76,488

Phase: 3

**Sponsor:** Ultragenyx Pharmaceutical Inc.

60 Leveroni Court

Novato, CA, USA 94949

**Author:** Ph.D.

Manager, Biostatistics, Biometrics

**Date:** 15DEC2016

Version Number: 1.0



## **Table of Contents**

| 1 | INTRODUCTION | | |
|---|---|---|---|
| 2 | STU | DY OBJECTIVES | 9 |
| | 2.1 | Primary Efficacy Objective | 9 |
| | 2.2 | Secondary Efficacy Objectives | 9 |
| | 2.3 | Exploratory Efficacy Objectives | 9 |
| | 2.4 | Pharmacokinetics Objective. | 9 |
| | 2.5 | Safety Objective | 9 |
| 3 | STU | DY DESIGN | 10 |
| | 3.1 | Overall Study Design and Plan | 10 |
| | 3.2 | Blinding and Randomization Methods | 11 |
| | 3.3 | Stratification Factors | 11 |
| | 3.4 | Determination of Sample Size | 11 |
| | 3.5 | Primary and Final Analyses | 11 |
| | 3.6 | Data Monitoring Committee | 12 |
| 4 | STU | DY CLINICAL OUTCOMES AND COVARIATES | 13 |
| | 4.1 | Primay Efficacy Endpoint | 13 |
| | 4.2 | Key Secondary Efficacy Endpoint | 13 |
| | 4.3 | Secondary Efficacy Endpoints | 13 |
| | 4.4 | Exploratory Efficacy Endpoints | 14 |
| | 4.5 | PK Endpoints | 14 |
| | 4.6 | Safety Endpoints | 14 |
| 5 | DEFINITIONS AND DERIVED EFFICACY VARIABLES | | |
| | 5.1 | Baseline | 16 |
| | 5.2 | Duration of Exposure | 16 |
| | 5.3 | Study Day | 16 |
| | 5.4 | Fractional Excretion of Phosphorus | 16 |



| | 5.5 | Iliac C | rest Bone Biopsy | 16 |
|---|---|---|---|---|
| | 5.6 | Brief P | ain Inventory | 17 |
| | 5.7 | Brief F | atigue Inventory | 17 |
| | 5.8 | Targete | ed Radiography and Skeletal Survey | 17 |
| | 5.9 | Time-A | Adjusted Area Under the Curve (AUC) | 18 |
| | 5.10 | Advers | ee Events To Monitor | 19 |
| | 5.11 | Prior m | nedication and Concomitant medication | 19 |
| 6 | ANA | ALYSIS | POPULATIONS | 20 |
| | 6.1 | Primar | y Analysis Set | 20 |
| | 6.2 | Full A | nalysis Set | 20 |
| | 6.3 | Safety | Analysis Set | 20 |
| | 6.4 | Treatm | ent Extension Analysis Set | 20 |
| | 6.5 | Pharma | acokinetics Analysis Set | 20 |
| 7 | DA | ΓA SCR | EENING AND ACCEPTANCE | 21 |
| | 7.1 | Handli | ng of Missing and Incomplete Data | 21 |
| | | 7.1.1 | Non-Responder Imputation | 21 |
| | | 7.1.2 | Missing Date Information for Adverse Events and Concomitant Medications | 21 |
| | | 7.1.3 | Missing Causal Relationship to Investigational Product for Adverse Events | 22 |
| | | 7.1.4 | Missing Data in Bone Biopsy Parameter MLt | 22 |
| | 7.2 | Unsche | eduled or Early Termination Visits | 22 |
| | 7.3 | Softwa | re | 23 |
| 8 | STA | TISTIC | AL METHODS OF ANALYSIS | 24 |
| | 8.1 | Genera | l Principles | 24 |
| | 8.2 | Subjec | t Accountability | 24 |
| | 8.3 | Protoco | ol Deviations | 24 |
| | 8.4 | Demog | graphics and Baseline Characteristics | 24 |



| | 8.5 | Disease | e Characteristics and Medical History | 25 |
|---|---|---|---|---|
| | | 8.5.1 | Medical History / XLH Medical History | 25 |
| | | 8.5.2 | XLH Treatment History | 25 |
| | 8.6 | 6 Efficacy Analysis | | |
| | | 8.6.1 | Primary Efficacy Endpoint | 25 |
| | | 8.6.2 | Key Secondary Efficacy Endpoint | 25 |
| | | 8.6.3 | Secondary Efficacy Endpoints | 26 |
| | | 8.6.4 | Exploratory Efficacy Endpoints | 27 |
| | 8.7 | PK An | alysis | 27 |
| | 8.8 | Genera | al Safety Analysis | 28 |
| | | 8.8.1 | Dosing Summary | 28 |
| | | 8.8.2 | Adverse Events | 28 |
| | | 8.8.3 | Prior and Concomitant Medications | 29 |
| | | 8.8.4 | Safety Lab Parameters | 29 |
| | | 8.8.5 | HAHA | 29 |
| | | 8.8.6 | Physical Examination | 29 |
| | | 8.8.7 | Pregnancy Test | 30 |
| | | 8.8.8 | Vital Signs | 30 |
| | 8.9 | Ectopic | c Mineralization Safety Analysis | 30 |
| | | 8.9.1 | Renal Ultrasound | 30 |
| | | 8.9.2 | ECG | 30 |
| | | 8.9.3 | ЕСНО | 31 |
| 9 | REF | ERENC | CES | 32 |
| 10 | APP | ENDIC | ES | 33 |
| | Appendix 1: Summary of Efficacy Endpoint and Analysis | | | |
| | Appendix 2: Brief Pain Inventory | | | |
| | Appendix 3: Brief Fatigue Inventory | | | |



| Appendix 4: Events to Monitor | 38 |
|--------------------------------|----|
| Appendix 5: Schedule of Events | 48 |



### **ABBREVIATIONS**

1,25[OH]<sub>2</sub>D 1,25-dihydroxyvitamin D

25(OH)D 25-hydroxy vitamin D

6MWT 6-Minute Walk Test

AE Adverse event

ALP Alkaline phosphatase
AUC Area under the curve

BALP Bone-specific alkaline phosphatase

BFI Brief fatigue inventory

BFR Bone formation rate

BPI Brief Pain Inventory

CFB Change from Baseline

CTCAE Common Terminology Criteria for Adverse Events

CTx Carboxy terminal cross-linked telopeptide of type I collagen

ECG Electrocardiogram

ECHO Echocardiogram

eGFR Estimated glomerular filtration rate

FGF23 Fibroblast growth factor 23

GEE Generalized Estimating Equation

GFR Glomerular filtration rate

HAHA Human anti-human antibody

iPTH Intact parathyroid hormone

ISR Injection site reactions

KRN23 Investigational product, an anti-FGF23 antibody

LVH Left ventricular hypertrophy

mAb Monoclonal antibody

MAR Mineral apposition rate

MLt Mineralization lag time



MedDRA Medical Dictionary for Regulatory Activities

MS/BS Mineralization surface/bone surface

OS/BS Osteoid surface/bone surface

O.Th Osteoid thickness

OV/BV Osteoid volume/bone volume

P1NP Procollagen type 1 N-propeptide

PD Pharmacodynamics

PHEX Phosphate-regulating gene with Homologies to Endopeptidases on the X-

chromosome

PK Pharmacokinetics

QTc Corrected QT interval

SAE Serious adverse event

SC Subcutaneous

SMQ Standardised MedDRA Query

TEAE Treatment-emergent adverse event

TmP/GFR Ratio of renal tubular maximum phosphate reabsorption rate to glomerular

filtration rate

TRP Tubular reabsorption of phosphate

WHO World Health Organization

XLH X-Linked Hypophosphatemia



## 1 INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide details of the statistical analyses planned for data collected under Ultragenyx Pharmaceutical Inc. Protocol UX023-CL304 titled "An Open-Label, Single-Arm, Phase 3 Study to Evaluate the Effects of KRN23 on Osteomalacia in Adults with X-linked Hypophosphatemia (XLH)." This SAP covers the original protocol and its two amendments, the latest of which was dated 07October 2016. Since the study protocol is a companion document to this SAP, aspects in the protocol unrelated to statistical issues (e.g., patient eligibility criteria and descriptions of clinical materials) are not repeated here. For all statistical matters, this SAP takes priority over any related statements on statistical matters within the protocol in the event there are any inconsistencies.



### 2 STUDY OBJECTIVES

### 2.1 Primary Efficacy Objective

Establish the effect of KRN23 treatment on improvement in XLH-associated osteomalacia as determined by osteoid volume (osteoid volume/bone volume, OV/BV)

### 2.2 Secondary Efficacy Objectives

The key secondary efficacy objective is to establish the effect of KRN23 treatment on increasing serum phosphorus levels in adults with XLH

Other secondary efficacy objectives are to establish the effect of KRN23 treatment in adults with XLH on:

- Changes from baseline in additional histomorphometric parameters including osteoid thickness (O.Th), osteoid surface/bone surface (OS/BS), and mineralization lag time (MLt)
- Changes from baseline in parameters of bone mineralization including mineral apposition rate (MAR), mineralizing surface (MS/BS), bone formation rate (BFR), and others
- Additional pharmacodynamics (PD) markers reflecting the status of phosphorus homeostasis and renal function
- Bone remodeling as assessed by bone turnover markers

### 2.3 Exploratory Efficacy Objectives

- Examine the effect of KRN23 treatment in adults with XLH on pseudofracture healing
- Patient reported outcomes (PROs) assessing skeletal pain and fatigue

### 2.4 Pharmacokinetics Objective

Assess the PK of KRN23 throughout the dosing cycle following the first doses and steady state

### 2.5 Safety Objective

Establish the safety and tolerability profile of KRN23 in the treatment of adults with XLH including adverse events (AEs), ectopic mineralization risk, cardiovascular effects, and immunogenicity profile



### 3 STUDY DESIGN

### 3.1 Overall Study Design and Plan

This is a Phase 3 open-label, single-arm, multicenter study to establish the effects of KRN23 on bone quality and osteomalacia associated with XLH. A total of 14 adult subjects with a diagnosis of XLH supported by typical clinical and biochemical features who have not received oral phosphate and vitamin D therapy in the past two years have been enrolled. To ensure a level of gender balance, at least 3 subjects of each sex have been enrolled. Iliac crest bone biopsies will be performed at baseline and 48 weeks. Baseline histologic and histomorphometric assessments of the bone biopsy specimens will be performed as each biopsy is completed to assess sample quality and confirm the presence of osteomalacia in at least 8 subjects. If a subject is determined not to have osteomalacia at the time of the initial biopsy, that subject will continue on study but will not undergo the second bone biopsy procedure at Week 48. All other assessments will be completed as scheduled. The goal of the study is to assess changes in bone quality. Histologic and histomorphometric evaluation of iliac crest bone biopsies will be supported by changes in serum phosphorus and biochemical markers of bone turnover and additional PD markers associated with FGF23-mediated processes. Pseudofractures and PROs will provide additional information on KRN23 efficacy. Safety, immunogenicity, and PK of KRN23 will also be evaluated.

KRN23 will be administered via subcutaneous (SC) injections monthly (Q4W, 28 days) for 48 weeks. Subjects who complete the 48 weeks of the Open-Label Treatment Period will then continue into an additional 48-week Treatment Extension Period. A Safety Follow-up Phone Call will be conducted 12 weeks (± 5 days) after the last dose of study drug.

All subjects will receive 1.0 mg/kg KRN23 monthly (Q4W, 28 days), rounded to the nearest 10 mg. The amount of drug administered will be calculated based on baseline weight and a 1.0 mg/kg KRN23 dose level (rounded to the nearest 10 mg) up to a maximum dose of 90 mg. The dose will remain fixed for the duration of the study, provided serum phosphorous levels do not exceed 5.0 mg/dL (1.61 mmol/L) at any time or 4.5 mg/dL (1.45 mmol/L) on two occasions. The dose will be recalculated if body weight changes by more than 20% from the baseline measurement.

Subjects will receive study drug via SC injection to the abdomen, upper arms, or thighs; the injection site will be rotated with each injection. No more than 1.5 mL may be administered to a single injection site. If the dose requires more than 1.5 mL, multiple injections must be administered, each at a different injection site.

If serum phosphorus increases above 5.0 mg/dL (1.61 mmol/L) at any time the actual dose will be decreased by half. If serum phosphorous increases above the ULN (4.5 mg/dL; 1.45 mmol/L) but does not exceed 5.0 mg/dL (1.61 mmol/L), the dose will be adjusted only if a second serum phosphorus result exceeds the ULN. Following a downward dose adjustment, the investigator together with the medical monitor should determine how and when to dose titrate up. Unscheduled serum phosphorus assessments may be necessary.



Based on the totality of the data from studies INT-001 and INT-002 over a period of 16 months in which most subjects were treated with 1.0 mg/kg KRN23 and no subject experienced an elevation of serum phosphorus that approached the 4.5 mg/dL (1.45 mmol/L) threshold, it is considered unlikely that dose adjustment will be necessary.

A complete schedule of events is included in Appendix 5.

## 3.2 Blinding and Randomization Methods

All subjects receive KRN23 on an open-label basis. Blinding and randomization are not applicable to this study design.

### 3.3 Stratification Factors

Not applicable.

## 3.4 Determination of Sample Size

The study will enroll approximately 14 adult subjects with XLH; baseline histologic and histomorphometric assessments of the bone biopsy specimens will be performed as each biopsy is completed to assess sample quality and confirm the presence of osteomalacia in at least 8 subjects. To ensure a level of gender balance, at least 3 subjects of each sex will be enrolled. At least 6 paired biopsy specimens are expected at the end of the study. A reduction in excess osteoid is expected to be shown in all subjects with paired biopsies with an estimated reduction from baseline in osteoid thickness. The sample size and study duration are believed to be sufficient to enable characterization of KRN23 effects on bone tissue and skeletal health.

Information will be used to support the findings of UX023-CL303 study which is a larger Phase 3 confirmatory efficacy and safety study, where it is adequately powered to evaluate increases in serum phosphorus levels across the entire dosing interval and to describe the treatment effect on select patient reported outcomes.

### 3.5 Primary and Final Analyses

The primary efficacy analysis will be performed after all subjects have completed Week 48 or discontinued from the study prior to week 48 and completed the post-baseline Bone Biopsy test for those who has been determined to have the osteomalacia at the baseline.

The final analysis will be performed after all subjects have completed the Week 96 assessments and the Safety Follow-up or discontinued from the study.

Administrative analyses during the Open Label Treatment Period and Treatment Extension Periods may be performed to support regulatory activities.



## 3.6 Data Monitoring Committee

An independent DMC that includes two clinicians with expertise in metabolic bone disease and one statistician will act in an advisory capacity to monitor subject safety on a routine basis throughout the trial. A review of safety data will be conducted by the DMC periodically. Ad hoc meetings will be held if indicated based on observed events. The roles and responsibilities of the DMC will be defined in the DMC Charter.



### 4 STUDY CLINICAL OUTCOMES AND COVARIATES

### 4.1 Primay Efficacy Endpoint

The primary endpoint is the percent change from baseline in osteoid volume/bone volume (OV/BV) at Week 48 based on analysis of iliac crest bone biopsies

## 4.2 Key Secondary Efficacy Endpoint

The key secondary efficacy endpoint is the proportion of subjects achieving mean serum phosphorus levels above the lower limit of normal (LLN; 2.5 mg/dL [0.81 mmol/L]) at the mid-point of the dose interval (i.e., Weeks 2, 6, 14, and 22), as averaged across dose cycles between baseline and Week 24.

## 4.3 Secondary Efficacy Endpoints

The secondary efficacy endpoints will compare the effects of treatment with KRN23 on the following:

- Percent changes from baseline in additional histomorphometric parameters including osteoid thickness (O.Th), osteoid surface/bone surface (OS/BS), and mineralization lag time (MLt) at Week 48
- Changes from baseline in MAR, MS/BS, BFR and additional measures of bone formation and remodeling at Week 48
- Additional measures to assess serum phosphorus levels between baseline and Week 24 include:
  - O Proportion of subjects achieving mean serum phosphorus levels above the LLN (2.5 mg/dL [0.81 mmol/L] at the end of the dosing cycle (4 weeks after dosing), as averaged across dose cycles
  - Mid-point of dosing cycle: mean change from baseline, and percent change from baseline averaged across dose cycles
  - End of dosing cycle: mean change from baseline, and percent change from baseline averaged across dose cycles
  - o Cumulative exposure: time-adjusted area under the curve (AUC)
- Change from baseline over time in serum phosphorus, serum intact FGF23, serum 1,25(OH)<sub>2</sub>D, urinary phosphorus, ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR), tubular reabsorption of phosphate (TRP), and fractional excretion of phosphorus (FEP)



• Change and percent change from baseline over time in serum bone turnover markers, including procollagen type 1 N-propeptide (P1NP), carboxy-terminal cross-linked telopeptide of type I collagen (CTx), and bone-specific alkaline phosphatase (BALP)

## 4.4 Exploratory Efficacy Endpoints

The following exploratory efficacy endpoints will be examined:

- The number of active pseudofractures as defined by skeletal survey at baseline and the number and percentage of the baseline active pseudofractures which healed, partially healed, were unchanged or worsened at post-baseline visits
- The number of subjects with baseline active pseudofractures and the number of those subjects who have changes from baseline to healed, partially healed, unchanged and worsened at post-baseline visits
- Change from baseline over time in Brief Pain Inventory (BPI) Q3 Worst Pain
- Change from baseline over time in BPI Pain Severity Score
- Change from baseline over time in Pain Interference scores
- Change from baseline over time in Brief Fatigue Inventory (BFI) Q3 Worst Fatigue scores
- Change from baseline over time in BFI Global Fatigue Score, calculated by averaging all 9 items on the BFI

## 4.5 PK Endpoints

Serum KRN23 concentrations will be obtained from all subjects at time points reflecting peak and trough drug concentration.

### 4.6 Safety Endpoints

Safety will be evaluated by the incidence, frequency and severity of AEs and serious adverse events (SAEs), including clinically significant changes from baseline to scheduled time points in the following safety variables:

General safety variables include:

- Vital signs and weight
- Physical examinations
- Estimated glomerular filtration rate (eGFR)



- Chemistry, hematology, and urinalysis, including additional KRN23/XLH biochemical parameters of interest (creatinine, calcium, and intact parathyroid hormone [iPTH])
- Immunogenicity (human anti-human antibodies; HAHA)
- Concomitant medications

Ectopic Mineralization Safety Assessments:

- Renal ultrasound
- Echocardiogram (ECHO) and electrocardiogram (ECG)



### 5 DEFINITIONS AND DERIVED EFFICACY VARIABLES

#### 5.1 Baseline

Baseline is defined as the last non-missing measurement taken prior to or on the first dose of Investigational Product (IP) administered in the study.

## 5.2 **Duration of Exposure**

Duration of exposure to IP in days is defined as the following:

For the primary analysis or other specified analysis before final analysis,

- The date at milestone visit (e.g. week 48) first date of IP + 1 day for the subjects completing the corresponding milestone visit
- Last date of IP first date of IP + 28 days for the subjects early discontinued

For final analysis:

• Last date of IP – first date of IP + 28 days

## 5.3 Study Day

Study Day 1 is the first date of IP.

- For visit date that is after Study Day 1, Study Day is calculated as the visit date the first date of IP +1.
- For visit date that is prior to Study Day 1, Study Day is calculated as the first date of IP the visit date.

### 5.4 Fractional Excretion of Phosphorus

Fractional excretion of phosphorus (FEP) is defined as 100%\*(2-hour urine phosphorus\*serum creatinine)/(2-hour urine creatinine \* serum phosphorus).

### 5.5 Iliac Crest Bone Biopsy

A bone biopsy of the iliac crest will be performed to assess OV/BV, O.Th, OS/BS, MLt as well as other parameters. Subjects will receive two courses of tetracycline (or demeclocycline) label prior to biopsy associated with the Baseline and Week 48 (or Early Termination if it occurs between the Week 24 and Week 48) visits. Bone biopsy of the trans-iliac crest will be performed by a physician trained and experienced in the procedure. Baseline bone biopsies will be qualitatively analyzed in real time to assess the presence of osteomalacia. If a subject is determined not to have osteomalacia at the time of the initial



biopsy, that subject will continue on study but will not undergo the second bone biopsy at Week 48/ET.

Primary and secondary efficacy endpoints derived from these assessments are provided in Section 8.8.

## 5.6 Brief Pain Inventory

The short-form Brief Pain Inventory (BPI) is an 11-question, self-reported, pain-specific questionnaire with a recall period of 24 hours that may allow a detailed characterization of the pain experienced by patients with XLH. The BPI will be administered at pre- and post-treatment time points as indicated in the Schedule of Events (Appendix 2) to assess pain severity and the impact of pain on daily functioning as measured by subject self-report.

The BPI endpoints to be analyzed are as follows:

- Worst pain, defined as the answer to question 3 (pain at its worst in the last 24 hours)
- Pain severity, defined as the average of questions 3 through 6
- Pain interference, defined as the average of questions 9A through 9G regarding the extent to which pain interfered with daily activities in the last 24 hours.

## 5.7 Brief Fatigue Inventory

The Brief Fatigue Inventory (BFI) is a self-reported questionnaire consisting of 9 items related to fatigue that are rated on a 0 to 10 numerical rating scale with a recall period of 24 hours. As with the BPI, two dimensions are measured: fatigue and the interference of fatigue on daily life (activity, mood, walking ability, work, relations with others, and enjoyment of life). The BFI will be administered at pre- and post-treatment time points as indicated in the Schedule of Events (Appendix 3) to assess fatigue severity and the impact of fatigue on daily functioning as measured by subject self-report.

The BFI endpoints to be analyzed are as follows:

- Worst fatigue, defined as the answer to question 3 (fatigue at its worst in the last 24 hours)
- BFI Global Fatigue score, defined as the average of all 9 items (questions 1 through 3 and questions 4A through 4F) on the BFI as recorded on the day of the study visit.

### 5.8 Targeted Radiography and Skeletal Survey

A radiographic skeletal survey will be conducted at baseline to assess healing or resolution of current pseudofractures, determine areas of osteomalacia and enthesopathy, and identify the number of pre-existing fractures/pseudofractures. Standard radiographs will be obtained of the chest, lateral spine, right and left hand/wrist, right and left humerus, right and left radius/ulna, right and left femur/pelvis, right and left tibia/fibula, and right and left foot.

Study Number: UX023-CL304

Statistical Analysis Plan 15DEC 2016, Version 1.0



During the 48-week long Open-Label Treatment Period, targeted radiography at locations identified by the skeletal survey will be taken at Weeks 12, 24, 36, and 48 to monitor frequency and healing of pseudofractures. During the Treatment Extension Period, targeted radiographs will only be taken at clinic visits following newly diagnosed fractures.

Post-baseline radiographs will be compared to baseline radiographs using a pre-defined list of abnormalities by a trained central reader who is blinded to subject data. Existing and new pseudofractures will be graded as not healed, partially healed, or fully healed.

## 5.9 Time-Adjusted Area Under the Curve (AUC)

The trapezoidal rule is a numerical method that approximates the value of a definite integral.

$$\int_{a}^{b} f(x) dx$$

Response versus time AUCs will be calculated using the trapezoidal rule. The formula for the area of a trapezoid is

$$Area = w\left(\frac{h_1 + h_2}{2}\right)$$

where w is the width of the trapezoid and h1 and h2 are the two heights as shown below



Each pair of consecutive response assessment times  $t_1$  and  $t_2$  form the width of a trapezoid with  $w_1 = t_2 - t_1$ . The heights  $h_1$  and  $h_2$  are the response values at times  $t_1$  and  $t_2$ , respectively. AUC is the sum of trapezoidal areas across specified time point.

$$\int_{a}^{b} f(x)dx \approx w_{1}\left(\frac{h_{1}+h_{2}}{2}\right) + w_{2}\left(\frac{h_{2}+h_{3}}{2}\right) + \dots + w_{n-1}\left(\frac{h_{n-1}+h_{n}}{2}\right)$$

AUC values can be normalized to time-adjusted AUCs by dividing AUC by the duration of time included in AUC calculation.

Time-Adjusted AUC = 
$$\frac{AUC}{\sum w_i}$$



### 5.10 Adverse Events To Monitor

**Injection Site Reaction (ISR)**: Defined by preferred terms under the Medical Dictionary for Regulatory Activities (MedDRA) high-level term (HLT) "Injection site reaction".

**Immunogenicity AE**: Defined using relevant PTs in the narrow SMQs for "Hypersensitivity".

**Hyperphosphataemia AE**: Defined by using PTs: "Hyperphosphataemia", "Blood phosphorus increased".

**Ectopic mineralization related AE**: There is no available SMQ. Ectopic mineralization related AE is defined using a MedDRA search of 'calcification'.

**Restless leg syndrome AE**:. Defined by PTs "Restless legs syndrome", "Restlessness", "Akathisia", "Sensory disturbance", "Psychomotor hyperactivity", "Limb discomfort", "Neuromuscular pain", "Formication".

See search criteria in Appendix 4.

### 5.11 Prior medication and Concomitant medication

Prior medication is defined as any medications start before the date of the first dose of IP.

Concomitant medication is defined as any medications that start before, on, or after the first dose of IP and continue into the treatment period.



### 6 ANALYSIS POPULATIONS

### 6.1 Primary Analysis Set

The primary analysis set will include enrolled subjects with baseline and follow-up (Week 48/ET) bone biopsy data.

## 6.2 Full Analysis Set

The full analysis set for efficacy is defined as all enrolled subjects who receive at least one dose of study drug. This analysis set will be used for the analyses of efficacy endpoints.

### 6.3 Safety Analysis Set

The safety analysis set consists of all enrolled subjects who receive at least one dose of study drug. This analysis set will be used for the analyses of all safety endpoints.

### 6.4 Treatment Extension Analysis Set

The treatment extension analysis set consists of all enrolled subjects who continued after the Open-Label Treatment Period and received at least one dose during the Treatment Extension Period. This analysis set will be used for the analyses of efficacy and safety endpoints after Week 48 analysis in additional to the full analysis set and safety analysis set.

## 6.5 Pharmacokinetics Analysis Set

The pharmacokinetics (PK) analysis set is the subset of subjects in the Safety analysis set who have at least 1 evaluable KRN23 concentration. The PK analysis set will be used for the analysis of the PK endpoints at each specific analysis milestone.



### 7 DATA SCREENING AND ACCEPTANCE

## 7.1 Handling of Missing and Incomplete Data

Missing clinical outcome data can occur for multiple reasons, including missed subject visits and measures with missing item scores. Missing and incomplete data will be identified through a review of tables and listings for this study. Missing and incomplete data will be identified for investigation, and possible resolution, by Data Management prior to the study database lock.

For all analyses, missing data will be treated as missing, unless otherwise specified. When a change from baseline is assessed, only subjects with a baseline and at least one post-baseline measurement will be included in the analysis.

## 7.1.1 Non-Responder Imputation

If no serum data is available to evaluate the key secondary endpoint, the subject will be considered as not achieving a serum phosphorus level above the LLN.

### 7.1.2 Missing Date Information for Adverse Events and Concomitant Medications

The following conventions will be used to impute missing portions of dates for adverse events and concomitant medications.

### Missing Start Dates

- If the day is unknown, then:
  - o If the month and year match the first dose of IP start date month and year in this study, then impute the day of the first dose date.
  - Otherwise, assign the first day of the month.
- If the month is unknown, then:
  - o If the year matches the year of the first dose of investigational product date in this study, then impute the month and day of the first dose date in this study.
  - o Otherwise, assign 'January'
- If the year is unknown, then the date will not be imputed and will be assigned a missing value.

## Missing Stop Dates

- If the day is unknown, then assign the last day of the month.
- If the month is unknown, then assign 'December.'
- If the year is unknown, then the date will not be imputed and will be assigned a missing value.



• If the resulting end date is after the date of study completion / discontinuation, set the imputed end date as the date of study completion / discontinuation.

## 7.1.3 Missing Causal Relationship to Investigational Product for Adverse Events

If the causal relationship to the investigational product is missing for an AE that started on or after the date of the first dose of double-blind investigational product, a causality of yes will be assigned. The imputed values for causal relationship to investigational product will be used for the incidence summary; the values will be shown as missing in the data listings.

## 7.1.4 Missing Data in Bone Biopsy Parameter MLt

1. If the MLt data is missing due to low quality of the bone biopsy sample (i.e. no bone biopsy parameters are available for that sample), the MLt parameter is set to missing for the sample. If the MLt data is missing due to very little label uptake because of the mineralization defect (i.e. there is at least one bone biopsy parameter available for that sample), the MLt will be imputed as O.Th/(MAR\*MS/OS), where MAR is imputed as 0.3 μm/day, using O.Th, MS and OS from the same visit of the same subject (Dempster et al. 2013). If any of O.Th, MS or OS at that visit for the subject is missing, MLt will be set as missing.

## 7.2 Unscheduled or Early Termination Visits

For an unscheduled visit occurring after the first dose date of IP, the unscheduled visit will be mapped into the closest post-baseline study scheduled visit for the assessment based on the study day of the unscheduled visit, and the target study day of the scheduled visit of the assessment in the protocol. If the unscheduled visit has the equal distance to the 2 study scheduled visits, it will be mapped to the later one.

The unscheduled visit will be only mapped to the study visit within each study period during which it occurs. If an unscheduled visit occurs during the Open-Label Treatment Period (from the first dose date to the dose date at week 48), it should be mapped to the study visit in the Open-Label Treatment Period. If an unscheduled visit occurs after the dose date at week 48 and in the Treatment Extension Period, it should be mapped to the study visit in the Treatment Extension Period.

When there is more than one measurement mapped to the same scheduled visit (including the original measurement taken from the scheduled visit), the measurement taken on the scheduled visit will be used if it is not missing, otherwise the one closest to the target day will be used. If more than one visit has the equal distance to the target day then the later one will be used. If more than one measurement is collected on the same day, use the time or the sequence number to select the latest record. For listings and shift tables, all data points will be included.

Early termination visit will follow the same rule for unscheduled visit as described above.



The bone biopsy taken in the early termination visit will not be mapped to the study scheduled visit as the bone biopsy will be only taken either on week 48 or at the early termination visit post-baseline used in the analysis.

### 7.3 Software

SAS® software version 9.4 or higher will be used to perform most or all statistical analyses.



### 8 STATISTICAL METHODS OF ANALYSIS

### 8.1 General Principles

The statistical analyses will be reported using summary tables, figures, and data listings. Statistical tests will be 2-sided at the alpha=0.05 significance level and 2-sided 95% confidence interval will be used. All p-values will be presented as nominal p-values. No adjustment on multiplicity will be made. Continuous variables will be summarized by number of subjects, mean, standard deviation (SD), standard error (SE), median, Q1, Q3, minimum, and maximum. Categorical variables will be summarized by number and percentages of subjects. No imputation on missing data will be made, unless stated otherwise.

When the sample size and number of observations allow, the change from baseline over time will be analyzed using a generalized estimation equation (GEE) model that includes time as the categorical variable and adjusted for baseline measurement. The covariance structure that will be used for the GEE model is compound symmetry which specifies constant variance for the assessments and constant covariance between the assessments over time. If the number of observations are insufficient for analyses using a GEE model, a t-test will be performed for continuous variables and a 95% confidence interval (CI) of the proportion will be provided for binary variables.

## 8.2 Subject Accountability

The number of subjects screened and enrolled, and the number and percentage of subjects in each analysis set will be summarized. The number and percentage of subjects who complete each treatment period and of subjects who prematurely discontinue during each treatment period and the study will be summarized. The reasons for study discontinuation will also be summarized. A subject disposition listing will be provided for individual subjects.

### **8.3** Protocol Deviations

Major and minor protocol deviations will be summarized separately by type for the Full analysis set. The protocol deviations recorded in the CRF will be listed.

#### 8.4 Demographics and Baseline Characteristics

Demographic characteristics and other baseline characteristics will be summarized descriptively for the Full Analysis Set and listed by subject including the following.

- Demographics: age, sex, race, ethnicity, height, weight, BMI, country and region
- Baseline Characteristics: baseline PD (serum phosphorus, etc.), renal ultrasound scores, baseline BPI-Q3, baseline skeletal survey radiographs measures, PHEX mutation



The summary of demographics and baseline characteristics will also be provided for the Primary Analysis Set when the number of subjects in the Primary Analysis Set is significantly fewer than the Full Analysis Set.

### 8.5 Disease Characteristics and Medical History

## 8.5.1 Medical History / XLH Medical History

Medical history will be summarized by body system for the Full Analysis set and will also be listed by subject. Fracture history will be summarized by reported term for the Full Analysis set and will also be listed by subject.

### 8.5.2 XLH Treatment History

The subjects' past XLH treatment with phosphates and vitamin D metabolites or analogs will be listed for the Full Analysis set if there is any reported XLH treatment history. For subjects receiving standard of care therapy for XLH (phosphate and/or vitamin D) the drug name, duration of treatment, dose and frequency of administration will be listed.

### 8.6 Efficacy Analysis

The primary efficacy analysis and other bone biopsy analysis (e.g. MAR, MS/BS, BFR, etc.) will be performed on the Primary Analysis set. All other efficacy analysis will be performed on the Full Analysis set at each milestone analysis. The treatment Extension Analysis Set might also be used for efficacy analysis at the final analysis.

### **8.6.1** Primary Efficacy Endpoint

The primary endpoint is the percent change from baseline at Week 48 in osteoid volume (osteoid volume/bone volume, OV/BV).

OV/BV at baseline, Week 48, both change from baseline, and percent change from baseline at Week 48 will be summarized. Change from baseline at Week 48 will be tested using a t-test if the normality assumption is valid. If the normal assumption is not met, a sign test will be used. The p-value from the statistical tests will be reported. A listing will be provided.

### 8.6.2 Key Secondary Efficacy Endpoint

The key secondary efficacy endpoint is the proportion of subjects achieving mean serum phosphorus levels above the LLN (2.5 mg/dL [0.81 mmol/L]) at the mid-point of the dose interval (i.e., Weeks 2, 6, 14, and 22), as averaged across dose cycles between baseline and Week 24.

The number and proportion of subjects achieving mean serum phosphorus levels above the LLN (2.5 mg/dL [0.81 mmol/L]) will be summarized and the two-sided 95% confidence interval will be provided for the proportion. The Wilson score method (Wilson 1927) will be



applied to estimate the confidence interval. The p-value for testing the proportion of subjects achieving the mean serum phosphorus levels above the LLN (2.5 mg/dL [0.81 mmol/L]) against 0% from the binomial test will also be provided.

### 8.6.3 Secondary Efficacy Endpoints

## 8.6.3.1 Additional bone biopsy endpoints

Analysis for the following parameters will use the same analysis method for the primary endpoint:

• Additional histomorphometric parameters – including osteoid thickness (O.Th), osteoid surface/bone surface (OS/BS), and mineralization lag time (MLt)

The observed, change from baseline, and percent change from baseline values over time for the following parameters will be summarized.

• MAR, MS/BS, BFR and additional measures of bone formation and remodeling

A listing of the bone biopsy parameters will be provided.

A sensitivity analysis for bone biopsy parameters based on the bone osteomalacia severity at baseline may also be explored. A shift analysis from baseline to post-baseline for the bone osteomalacia severity based on the category reported in the EDC may also be performed.

## 8.6.3.2 Key PD

Descriptive summaries of the following secondary PD endpoints will be provided.

- Proportion of subjects achieving mean serum phosphorus levels above the LLN (2.5 mg/dL [0.81 mmol/L]) at the end of the dosing cycle (4 weeks after dosing), as averaged across dose cycles between baseline and week 24.
- Mean change from baseline and percent change from baseline in serum phosphorus at each mid-point of dosing cycle, as averaged across dose cycles between baseline and week 24.
- Mean change from baseline and percent change from baseline in serum phosphorus at each end of dosing cycle, as averaged across dose cycles between baseline and week 24.
- Time-adjusted area under the curve (AUC) of serum phosphorus between baseline and week 24.

Observed values and change from baseline, serum intact FGF23, percent change from baseline over time in serum phosphorus, 1,25(OH)<sub>2</sub>D, and urinary phosphorus, TRP, TmP/GFR, and FEP will be summarized at each milestone analysis.



The change from baseline over time for key PD will be analyzed using the GEE model as described in Section 8.1, if the model converges.

A listing for the PD parameters will be provided.

Mean ( $\pm$ SE) PD-time plots may be presented for the PD parameters.

#### **8.6.3.3** Bone turnover markers

Observed values, change and percent change from baseline over time in serum ALP and biochemical markers of bone turnover, including BALP, CTx, and P1NP, will be summarized at each milestone analysis. A listing will be provided for the biochemical markers of bone turnover.

The change from baseline over time for biomarkers will also be analyzed using the GEE model as described in Section 8.1, if the model converges.

Correlations may be used to assess the relationship between bone turnover markers and selected histomorphometric indices.

### **8.6.4** Exploratory Efficacy Endpoints

The number of active (non-healed) pseudofractures and/or fractures as defined by skeletal survey at baseline and the number and percentage of the baseline active pseudofractures/fractures which healed, partially healed, were unchanged or worsened at post-baseline visits will be summarized. New active pseudofractures and/or fractures identified at post-baseline visits will also be summarized.

The number of the subjects with baseline active pseudofractures and/or fractures and the number of those subjects who have changes from baseline to healed, partially healed, unchanged and worsened at post-baseline visits will be summarized. The number of subjects with new active pseudofractures and/or fractures at post-baseline visits will also be summarized.

For BPI (worst pain, pain severity and pain interference), BFI (worst fatigue, and global fatigue score), the observed values, change from baseline over time will be summarized. The change from baseline over time will also be analyzed using the GEE model as described in Section 8.1, if the model converges. Listings for the patient-reported outcomes will be provided.

### 8.7 PK Analysis

All PK analyses will be performed for subjects in the PK Analysis set with evaluable serum PK samples. Serum KRN23 will be summarized descriptively at each time point.



## 8.8 General Safety Analysis

All safety analyses will be performed on the Safety Analysis set at each milestone analysis. The treatment Extension Analysis Set might also be used for safety analysis at the final analysis. General safety will include dosing summary, AEs, treatment related AEs, SAEs, events to monitor, prior and concomitant medication, laboratory measurements including chemistry, hematology, and urinalysis parameters, GFR, amylase, HAHA, pregnancy test and vital signs. No hypothesis testing is planned for safety data.

## **8.8.1 Dosing Summary**

The total dose administered and the subjects with dose adjustment and the reasons for dose adjustment will be summarized by treatment groups by visits for the safety analysis set.

#### **8.8.2** Adverse Events

Reported adverse event (AE) terms are coded to MedDRA (version 18.1). All reported events will appear in AE listings, however only TEAEs will be summarized. TEAEs are defined as AEs occurring or worsened in severity on or after the first dose date of IP.

The following AEs will be summarized at each milestone analysis:

- All TEAEs
- Related TEAEs
- TEAE by severity
- Events to monitor:
  - Injection site reactions
  - o Immunogenicity
  - o Hyperphosphataemia
  - o Ectopic mineralization
  - Restless legs syndrome
- Grade 3/4 TEAEs
- Serious TEAEs
- Serious related TEAEs
- TEAEs resulting in discontinuation
- Fatal TEAEs.

The incidence and frequency of AEs will be summarized by System Organ Class (SOC), Preferred Term (PT). Events to monitor will be summarized by PT. Injection site reactions (ISR) will be listed for PT, seriousness, severity, outcome, relationship to study drug, and onset time from IP administration.

Listings will be created for AEs which lead to death, discontinuation of treatment, and SAEs.



### 8.8.3 Prior and Concomitant Medications

Both prior and concomitant medications will be coded by drug name and therapeutic class using WHO Drug dictionary, version 2015 September or newer.

Prior medication will be summarized by therapeutic class and preferred term at week 48 analysis.

At each specific milestone analysis, concomitant medications will be summarized by therapeutic class and preferred term.

## 8.8.4 Safety Lab Parameters

The descriptive statistics will be provided for lab safety parameters (chemistry, hematology, and urinalysis parameters, serum 25(OH)D, FGF23, lipase, amylase, eGFR). Observed values and change from baseline will be presented.

In addition, a shift table will be provided for amylase. The following categories will be used for serum amylase:

- No Grade
- Grade 1: >ULN to 1.5 x ULR
- Grade 2: >1.5 to 2 x ULR
- Grade 3: >2 to 5 x ULR
- Grade 4: > 5 x ULR

Individual and mean (±SE) over time plots may be presented for selected safety lab parameters.

Listings of the lab safety parameters will be provided.

#### 8.8.5 HAHA

Antibody (human anti-human antibody [HAHA]) results will be summarized by the baseline and post-baseline testing results. Each subject positive for antibody will be listed with titer (if available), the cumulative dose of KRN23 up to the time of the positive antibody test, the time since the first exposure to KRN23, and the latest dose of KRN23 before the positive antibody test.

### 8.8.6 Physical Examination

Physical exam results will include the assessment of general appearance; head, eyes, ears, nose, and throat; the cardiovascular, dermatology, lymphatic, respiratory, gastrointestinal, musculoskeletal, genitourinary, neurological systems. All physical examination assessments will be listed.



## 8.8.7 Pregnancy Test

A subject level listing for pregnancy test results will be created for those who had a positive pregnancy test.

### 8.8.8 Vital Signs

Systolic blood pressure, diastolic blood pressure, temperature, respiratory rate and heart rate and their changes from baseline over time will be summarized. If the subject has taken 2 measurements of BP separated by 15 min at the same scheduled visit per the protocol amendment 1, the mean of the 2 measurements of the blood pressure at the visit will be used for analysis.

## 8.9 Ectopic Mineralization Safety Analysis

Ectopic mineralization safety data includes renal ultrasound, ECG, ECHO, serum calcium, phosphorus, intact parathyroid hormone (iPTH), urinary calcium and creatinine. The observed values and changes from baseline in the ectopic mineralization labs (serum calcium etc.) will be summarized. Listings containing the ectopic mineralization safety parameters will be provided.

#### 8.9.1 Renal Ultrasound

Renal ultrasound will be conducted with findings of nephrocalcinosis graded on a 5-point scale and by a central reader. These results will be summarized by time point. Furthermore, a grade shift table summarizing changes from baseline by time point will also be created.

The number and percentage of subjects with nephrolithiasis observed in the cortical collecting duct will be summarized by time point. A shift table summarizing changes from baseline by time point will be created.

A listing of renal ultrasound nephrocalcinosis scores, the presence or absence of nephrolithiasis in the cortical collecting duct and the radiologist's comments will also be provided.

#### 8.9.2 ECG

Summary statistics for the absolute measurements and changes from Baseline for selected ECG parameters including the following intervals: QT, QTcF - Fridericia's Correction Formula, the time elapsed from the onset of atrial depolarization to the onset of ventricular depolarization (PR), RR duration, and time elapsed for depolarization of the ventricles (QRS) will be provided.

ECG parameters will also be summarized by the maximum post-baseline value and maximum change from baseline using the following categories based on International Conference on Harmonisation (ICH) E14 (ICH 2005).



## Categories for ECG Results

| ECG<br>Parameter | Categories for Baseline and Maximum<br>Post-Baseline Value | Categories for Maximum Change from Baseline Value |
|---|---|---|
| QTcF | ≤450, >450-≤480, >480-≤500 and >500 msec | ≤30, >30-≤60 and >60 msec |

The normality or abnormality of the ECG tracing will be summarized using shift tables of numbers of subjects who have a normal/abnormal ECG tracing by visits.

### 8.9.3 ECHO

ECHO data will be centrally read to assess for evidence of ectopic mineralization in the heart and aorta and to evaluate for signs of LVH or cardiac dysfunction. Descriptive statistics for the various continuous ECHO measurements (e.g., left ventricular mass index, etc.) will be at the scheduled time points and will include the change from baseline value. The summary of the descriptive statistics will be displayed by visit. The categorical summaries for the subjects with change from baseline >=2 in ectopic mineralization score will be performed. Shift tables will be provided for categorical ECHO measurements (e.g. ectopic mineralization score, aortic and mitral valve regurgitation).

A listing of all ECHO parameters will also be created.



### 9 REFERENCES

Dempster, DW, Compston, JE, Drezner, MK, Glorieux, FH, Kanis, JA, Malluche, H, Meunier, PJ, Ott, SM, Recker, RR, and Parfitt, AM. 2013. "Standardized nomenclature, symbols, and units for bone histomorphometry: a 2012 update of the report of the ASBMR Histomorphometry Nomenclature Committee." *J Bone Miner Res* 28 (1):2-17.

ICH. The International Conference on Harmonisation. E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs. 2005.

Wilson, E. B. (1927). Probable inference, the law of succession, and statistical inference. Journal of the American Statistical Association 22: 209–212



## 10 APPENDICES

# **Appendix 1: Summary of Efficacy Endpoint and Analysis**

| Test /<br>Instrument | Endpoint | Туре | Time points for Assessment | Statistical Analysis |
|---|---|---|---|---|
| Bone Biopsy | The primary endpoint is the percent change from baseline in osteoid volume/bone volume (OV/BV) at Week 48 based on analysis of iliac crest bone biopsies. | Primary Efficacy Endpoints | Baseline, 48/ET | Descriptive Summary<br>and T-Test (or Sign<br>Test) |
| Serum Phosphorus | The proportion of subjects achieving mean serum phosphorus levels above 2.5 mg/dL at the mid-point of the dose interval as averaged across dose cycles between baseline and Week 24. | Key Secondary Efficacy<br>Endpoints | Screening, Baseline,<br>Week 1, 2, 4, 6,<br>12,14,20,21, 22,<br>24,28, 36, 48, 60, 70,<br>72, 84, 94, 96, ET. | Descriptive Summary<br>and Wilson Confidence<br>Interval |
| Bone Biopsy | Percent changes from baseline in additional histomorphometric parameters – including osteoid thickness (O.Th), osteoid surface/bone surface (OS/BS), and mineralization lag time (MLt) | Secondary Efficacy Endpoints | Baseline, 48/ET | Descriptive Summary<br>and T-Test (or Sign<br>Test) |
| Bone Biopsy | Changes from baseline in MAR, MS/BS,<br>BFR and additional measures of bone<br>formation and remodeling | Secondary Efficacy Endpoints | Baseline, 48/ET | Descriptive Summary |
| Serum Phosphorus | Proportion of subjects achieving mean serum phosphorus levels above 2.5 mg/dL at the end of the dosing cycle, as averaged across dose cycles | Secondary Efficacy Endpoints | Screening, Baseline,<br>Week 1, 2, 4, 6,<br>12,14,20,21, 22,<br>24,28, 36, 48, 60, 70, | Descriptive Summary |
| | Mid-point of dosing cycle: mean change from baseline and percent change from baseline averaged across dose cycles through Week 24 | Secondary Efficacy Endpoints | 72, 84, 94, 96, ET. | Descriptive Summary |
| | End of dosing cycle: mean change from baseline averaged across dose cycles | Secondary Efficacy Endpoints | | Descriptive Summary |
| | Cumulative exposure: Time Adjusted area under the curve (AUC) | Secondary Efficacy Endpoints | | Descriptive Summary |




| Test /<br>Instrument | Endpoint | Туре | Time points for Assessment | Statistical Analysis |
|---|---|---|---|---|
| PD | Change from baseline over time in serum intact FGF23, ALP, 1,25(OH)2D; and urinary phosphorus, TRP,TmP/GFR, and FEP | Secondary Efficacy Endpoints | Screening, Baseline,<br>Week 1, 2, 4,<br>12,20,21, 22, 24,36,<br>48, 60, 72, 84, 94, 96,<br>ET. | Descriptive Summary ,<br>GEE Model |
| Biomarker | Change and percent change from baseline over time in bone biomarker, including BALP, CTx, P1NP, and osteocalcin | Secondary Efficacy Endpoints | Baseline, week 12, 24, 48, 72, 96 and ET. | Descriptive Summary ,<br>GEE Model |
| X-Ray | Number of post-baseline healed, partial healed pseudofractures from baseline active pseudofractures; Number of subjects who have active pseudofractures at baseline and healed, partial healed post-baseline pseudofractures | Exploratory Efficacy Endpoints | Baseline, week 12, 24, 36, 48 and ET. | Descriptive Summary ,<br>GEE Model |
| ВРІ | Change from baseline in: Worst Pain Pain Severity Pain Interference | Exploratory Efficacy Endpoints | Screening, Baseline, week 12, 24, 36, 48, 72, 96 and ET. | Descriptive Summary ,<br>GEE Model |
| BFI | Change from Baseline in: Worst Fatigue Global Fatigue Score | Exploratory Efficacy Endpoints | Screening, Baseline, week 12, 24, 36, 48, 72, 96 and ET. | |




**Appendix 2: Brief Pain Inventory** 








**Appendix 3: Brief Fatigue Inventory** 





### **Appendix 4: Events to Monitor**

Injection site reactions: based on HLT "Injection site reaction"

| Category | PT |
|-------------------------|----------------------------------|
| Injection site reaction | Embolia cutis medicamentosa |
| Injection site reaction | Injected limb mobility decreased |
| Injection site reaction | Injection site abscess |
| Injection site reaction | Injection site abscess sterile |
| Injection site reaction | Injection site anaesthesia |
| Injection site reaction | Injection site atrophy |
| Injection site reaction | Injection site bruising |
| Injection site reaction | Injection site calcification |
| Injection site reaction | Injection site cellulitis |
| Injection site reaction | Injection site coldness |
| Injection site reaction | Injection site cyst |
| Injection site reaction | Injection site dermatitis |
| Injection site reaction | Injection site discharge |
| Injection site reaction | Injection site discolouration |
| Injection site reaction | Injection site discomfort |
| Injection site reaction | Injection site dryness |
| Injection site reaction | Injection site dysaesthesia |
| Injection site reaction | Injection site eczema |
| Injection site reaction | Injection site erosion |
| Injection site reaction | Injection site erythema |
| Injection site reaction | Injection site exfoliation |
| Injection site reaction | Injection site extravasation |
| Injection site reaction | Injection site fibrosis |
| Injection site reaction | Injection site granuloma |
| Injection site reaction | Injection site haematoma |
| Injection site reaction | Injection site haemorrhage |
| Injection site reaction | Injection site hyperaesthesia |
| Injection site reaction | Injection site hypersensitivity |
| Injection site reaction | Injection site hypertrichosis |
| Injection site reaction | Injection site hypertrophy |
| Injection site reaction | Injection site hypoaesthesia |
| Injection site reaction | Injection site induration |
| Injection site reaction | Injection site infection |
| Injection site reaction | Injection site inflammation |
| Injection site reaction | Injection site injury |
| Injection site reaction | Injection site irritation |
| Injection site reaction | Injection site ischaemia |
| Injection site reaction | Injection site joint discomfort |



| Category | PT |
|-------------------------|------------------------------------------|
| Injection site reaction | Injection site joint effusion |
| Injection site reaction | Injection site joint erythema |
| Injection site reaction | Injection site joint infection |
| Injection site reaction | Injection site joint inflammation |
| Injection site reaction | Injection site joint movement impairment |
| Injection site reaction | Injection site joint pain |
| Injection site reaction | Injection site joint swelling |
| Injection site reaction | Injection site joint warmth |
| Injection site reaction | Injection site laceration |
| Injection site reaction | Injection site lymphadenopathy |
| Injection site reaction | Injection site macule |
| Injection site reaction | Injection site mass |
| Injection site reaction | Injection site movement impairment |
| Injection site reaction | Injection site necrosis |
| Injection site reaction | Injection site nerve damage |
| Injection site reaction | Injection site nodule |
| Injection site reaction | Injection site oedema |
| Injection site reaction | Injection site pain |
| Injection site reaction | Injection site pallor |
| Injection site reaction | Injection site papule |
| Injection site reaction | Injection site paraesthesia |
| Injection site reaction | Injection site phlebitis |
| Injection site reaction | Injection site photosensitivity reaction |
| Injection site reaction | Injection site plaque |
| Injection site reaction | Injection site pruritus |
| Injection site reaction | Injection site pustule |
| Injection site reaction | Injection site rash |
| Injection site reaction | Injection site reaction |
| Injection site reaction | Injection site recall reaction |
| Injection site reaction | Injection site scab |
| Injection site reaction | Injection site scar |
| Injection site reaction | Injection site streaking |
| Injection site reaction | Injection site swelling |
| Injection site reaction | Injection site thrombosis |
| Injection site reaction | Injection site ulcer |
| Injection site reaction | Injection site urticaria |
| Injection site reaction | Injection site vasculitis |
| Injection site reaction | Injection site vesicles |
| Injection site reaction | Injection site warmth |
| Injection site reaction | Malabsorption from injection site |



Immunogenicity: based on relevant PTs in the narrow SMQs for "Hypersensitivity",

| Category | PT |
|------------------|--------------------------------------------|
| Hypersensitivity | Acute generalised exanthematous pustulosis |
| Hypersensitivity | Administration site dermatitis |
| Hypersensitivity | Administration site eczema |
| Hypersensitivity | Administration site hypersensitivity |
| Hypersensitivity | Administration site rash |
| Hypersensitivity | Administration site recall reaction |
| Hypersensitivity | Administration site urticaria |
| Hypersensitivity | Administration site vasculitis |
| Hypersensitivity | Allergic bronchitis |
| Hypersensitivity | Allergic colitis |
| Hypersensitivity | Allergic cough |
| Hypersensitivity | Allergic cystitis |
| Hypersensitivity | Allergic eosinophilia |
| Hypersensitivity | Allergic gastroenteritis |
| Hypersensitivity | Allergic granulomatous angiitis |
| Hypersensitivity | Allergic hepatitis |
| Hypersensitivity | Allergic keratitis |
| Hypersensitivity | Allergic myocarditis |
| Hypersensitivity | Allergic oedema |
| Hypersensitivity | Allergic otitis externa |
| Hypersensitivity | Allergic otitis media |
| Hypersensitivity | Allergic pharyngitis |
| Hypersensitivity | Allergic respiratory disease |
| Hypersensitivity | Allergic respiratory symptom |
| Hypersensitivity | Allergic sinusitis |
| Hypersensitivity | Allergic transfusion reaction |
| Hypersensitivity | Allergy alert test positive |
| Hypersensitivity | Allergy test positive |
| Hypersensitivity | Allergy to immunoglobulin therapy |
| Hypersensitivity | Allergy to vaccine |
| Hypersensitivity | Alveolitis allergic |
| Hypersensitivity | Anaphylactic reaction |
| Hypersensitivity | Anaphylactic shock |
| Hypersensitivity | Anaphylactic transfusion reaction |
| Hypersensitivity | Anaphylactoid reaction |
| Hypersensitivity | Anaphylactoid shock |
| Hypersensitivity | Anaphylaxis treatment |
| Hypersensitivity | Angioedema |



| Category | PT |
|------------------|----------------------------------------------------------|
| Hypersensitivity | Antiallergic therapy |
| Hypersensitivity | Antiendomysial antibody positive |
| Hypersensitivity | Anti-neutrophil cytoplasmic antibody positive vasculitis |
| Hypersensitivity | Application site dermatitis |
| Hypersensitivity | Application site eczema |
| Hypersensitivity | Application site hypersensitivity |
| Hypersensitivity | Application site rash |
| Hypersensitivity | Application site recall reaction |
| Hypersensitivity | Application site urticaria |
| Hypersensitivity | Application site vasculitis |
| Hypersensitivity | Arthritis allergic |
| Hypersensitivity | Atopy |
| Hypersensitivity | Blepharitis allergic |
| Hypersensitivity | Blood immunoglobulin E abnormal |
| Hypersensitivity | Blood immunoglobulin E increased |
| Hypersensitivity | Bromoderma |
| Hypersensitivity | Bronchospasm |
| Hypersensitivity | Catheter site dermatitis |
| Hypersensitivity | Catheter site eczema |
| Hypersensitivity | Catheter site hypersensitivity |
| Hypersensitivity | Catheter site rash |
| Hypersensitivity | Catheter site urticaria |
| Hypersensitivity | Catheter site vasculitis |
| Hypersensitivity | Chronic eosinophilic rhinosinusitis |
| Hypersensitivity | Chronic hyperplastic eosinophilic sinusitis |
| Hypersensitivity | Circulatory collapse |
| Hypersensitivity | Circumoral oedema |
| Hypersensitivity | Conjunctival oedema |
| Hypersensitivity | Conjunctivitis allergic |
| Hypersensitivity | Corneal oedema |
| Hypersensitivity | Cutaneous vasculitis |
| Hypersensitivity | Dennie-Morgan fold |
| Hypersensitivity | Dermatitis |
| Hypersensitivity | Dermatitis acneiform |
| Hypersensitivity | Dermatitis allergic |
| Hypersensitivity | Dermatitis atopic |
| Hypersensitivity | Dermatitis bullous |
| Hypersensitivity | Dermatitis contact |
| Hypersensitivity | Dermatitis exfoliative |
| Hypersensitivity | Dermatitis exfoliative generalised |



| Category | PT |
|------------------|-------------------------------------------------------|
| Hypersensitivity | Dermatitis herpetiformis |
| Hypersensitivity | Dermatitis infected |
| Hypersensitivity | Dermatitis psoriasiform |
| Hypersensitivity | Distributive shock |
| Hypersensitivity | Documented hypersensitivity to administered product |
| Hypersensitivity | Drug cross-reactivity |
| Hypersensitivity | Drug eruption |
| Hypersensitivity | Drug hypersensitivity |
| Hypersensitivity | Drug provocation test |
| Hypersensitivity | Drug reaction with eosinophilia and systemic symptoms |
| Hypersensitivity | Eczema |
| Hypersensitivity | Eczema infantile |
| Hypersensitivity | Eczema nummular |
| Hypersensitivity | Eczema vaccinatum |
| Hypersensitivity | Eczema vesicular |
| Hypersensitivity | Eczema weeping |
| Hypersensitivity | Encephalitis allergic |
| Hypersensitivity | Encephalopathy allergic |
| Hypersensitivity | Epidermal necrosis |
| Hypersensitivity | Epidermolysis |
| Hypersensitivity | Epidermolysis bullosa |
| Hypersensitivity | Epiglottic oedema |
| Hypersensitivity | Erythema multiforme |
| Hypersensitivity | Erythema nodosum |
| Hypersensitivity | Exfoliative rash |
| Hypersensitivity | Eye allergy |
| Hypersensitivity | Eye oedema |
| Hypersensitivity | Eye swelling |
| Hypersensitivity | Eyelid oedema |
| Hypersensitivity | Face oedema |
| Hypersensitivity | Giant papillary conjunctivitis |
| Hypersensitivity | Gingival oedema |
| Hypersensitivity | Gingival swelling |
| Hypersensitivity | Gleich's syndrome |
| Hypersensitivity | Haemorrhagic urticaria |
| Hypersensitivity | Hand dermatitis |
| Hypersensitivity | Henoch-Schonlein purpura |
| Hypersensitivity | Henoch-Schonlein purpura nephritis |
| Hypersensitivity | Hereditary angioedema |
| Hypersensitivity | Hypersensitivity |



| Category | PT |
|------------------|---------------------------------------|
| Hypersensitivity | Hypersensitivity vasculitis |
| Hypersensitivity | Idiopathic urticaria |
| Hypersensitivity | Immediate post-injection reaction |
| Hypersensitivity | Immune thrombocytopenic purpura |
| Hypersensitivity | Immune tolerance induction |
| Hypersensitivity | Infusion site dermatitis |
| Hypersensitivity | Infusion site eczema |
| Hypersensitivity | Infusion site hypersensitivity |
| Hypersensitivity | Infusion site rash |
| Hypersensitivity | Infusion site recall reaction |
| Hypersensitivity | Infusion site urticaria |
| Hypersensitivity | Infusion site vasculitis |
| Hypersensitivity | Injection site dermatitis |
| Hypersensitivity | Injection site eczema |
| Hypersensitivity | Injection site hypersensitivity |
| Hypersensitivity | Injection site rash |
| Hypersensitivity | Injection site recall reaction |
| Hypersensitivity | Injection site urticaria |
| Hypersensitivity | Injection site vasculitis |
| Hypersensitivity | Instillation site hypersensitivity |
| Hypersensitivity | Instillation site rash |
| Hypersensitivity | Instillation site urticaria |
| Hypersensitivity | Interstitial granulomatous dermatitis |
| Hypersensitivity | Intestinal angioedema |
| Hypersensitivity | Iodine allergy |
| Hypersensitivity | Kaposi's varicelliform eruption |
| Hypersensitivity | Kounis syndrome |
| Hypersensitivity | Laryngeal oedema |
| Hypersensitivity | Laryngitis allergic |
| Hypersensitivity | Laryngospasm |
| Hypersensitivity | Laryngotracheal oedema |
| Hypersensitivity | Limbal swelling |
| Hypersensitivity | Lip oedema |
| Hypersensitivity | Lip swelling |
| Hypersensitivity | Mast cell degranulation present |
| Hypersensitivity | Mouth swelling |
| Hypersensitivity | Mucocutaneous rash |
| Hypersensitivity | Multiple allergies |
| Hypersensitivity | Nephritis allergic |
| Hypersensitivity | Nikolsky's sign |



| Category | PT |
|------------------|-------------------------------------------------|
| Hypersensitivity | Nodular rash |
| Hypersensitivity | Oculomucocutaneous syndrome |
| Hypersensitivity | Oculorespiratory syndrome |
| Hypersensitivity | Oedema mouth |
| Hypersensitivity | Oral allergy syndrome |
| Hypersensitivity | Oropharyngeal blistering |
| Hypersensitivity | Oropharyngeal spasm |
| Hypersensitivity | Oropharyngeal swelling |
| Hypersensitivity | Palatal oedema |
| Hypersensitivity | Palatal swelling |
| Hypersensitivity | Palisaded neutrophilic granulomatous dermatitis |
| Hypersensitivity | Palpable purpura |
| Hypersensitivity | Pathergy reaction |
| Hypersensitivity | Periorbital oedema |
| Hypersensitivity | Pharyngeal oedema |
| Hypersensitivity | Pruritus allergic |
| Hypersensitivity | Radioallergosorbent test positive |
| Hypersensitivity | Rash |
| Hypersensitivity | Rash erythematous |
| Hypersensitivity | Rash follicular |
| Hypersensitivity | Rash generalised |
| Hypersensitivity | Rash macular |
| Hypersensitivity | Rash maculo-papular |
| Hypersensitivity | Rash maculovesicular |
| Hypersensitivity | Rash morbilliform |
| Hypersensitivity | Rash neonatal |
| Hypersensitivity | Rash papulosquamous |
| Hypersensitivity | Rash pruritic |
| Hypersensitivity | Rash pustular |
| Hypersensitivity | Rash rubelliform |
| Hypersensitivity | Rash scarlatiniform |
| Hypersensitivity | Rash vesicular |
| Hypersensitivity | Reaction to azo-dyes |
| Hypersensitivity | Reaction to colouring |
| Hypersensitivity | Reaction to drug excipients |
| Hypersensitivity | Reaction to preservatives |
| Hypersensitivity | Red man syndrome |
| Hypersensitivity | Rhinitis allergic |
| Hypersensitivity | Scleral oedema |
| Hypersensitivity | Scleritis allergic |



| Category | PT |
|------------------|-------------------------------------------|
| Hypersensitivity | Scrotal oedema |
| Hypersensitivity | Serum sickness |
| Hypersensitivity | Serum sickness-like reaction |
| Hypersensitivity | Shock |
| Hypersensitivity | Shock symptom |
| Hypersensitivity | Skin necrosis |
| Hypersensitivity | Skin reaction |
| Hypersensitivity | Skin test positive |
| Hypersensitivity | Solar urticaria |
| Hypersensitivity | Solvent sensitivity |
| Hypersensitivity | Stevens-Johnson syndrome |
| Hypersensitivity | Stoma site hypersensitivity |
| Hypersensitivity | Stoma site rash |
| Hypersensitivity | Swelling face |
| Hypersensitivity | Swollen tongue |
| Hypersensitivity | Tongue oedema |
| Hypersensitivity | Toxic epidermal necrolysis |
| Hypersensitivity | Toxic skin eruption |
| Hypersensitivity | Tracheal oedema |
| Hypersensitivity | Type I hypersensitivity |
| Hypersensitivity | Type II hypersensitivity |
| Hypersensitivity | Type III immune complex mediated reaction |
| Hypersensitivity | Type IV hypersensitivity reaction |
| Hypersensitivity | Urticaria |
| Hypersensitivity | Urticaria cholinergic |
| Hypersensitivity | Urticaria chronic |
| Hypersensitivity | Urticaria contact |
| Hypersensitivity | Urticaria papular |
| Hypersensitivity | Urticaria physical |
| Hypersensitivity | Urticaria pigmentosa |
| Hypersensitivity | Urticaria vesiculosa |
| Hypersensitivity | Vaginal exfoliation |
| Hypersensitivity | Vaginal ulceration |
| Hypersensitivity | Vasculitic rash |
| Hypersensitivity | Vessel puncture site rash |
| Hypersensitivity | Vulval ulceration |
| Hypersensitivity | Vulvovaginal rash |
| Hypersensitivity | Vulvovaginal ulceration |



Hyperphosphataemia: based on selected PTs below

| Category | PT |
|--------------------|----------------------------|
| Hyperphosphataemia | Hyperphosphataemia |
| Hyperphosphataemia | Blood phosphorus increased |

Ectopic mineralization: based on a MedDRA search of 'calcification'

| Category | PT |
|-----------------------|-----------------------------------|
| Ectopic calcification | Adrenal calcification |
| Ectopic calcification | Aortic calcification |
| Ectopic calcification | Aortic valve calcification |
| Ectopic calcification | Aortic valve sclerosis |
| Ectopic calcification | Articular calcification |
| Ectopic calcification | Bladder wall calcification |
| Ectopic calcification | Breast calcifications |
| Ectopic calcification | Bursa calcification |
| Ectopic calcification | Calcific deposits removal |
| Ectopic calcification | Calcification metastatic |
| Ectopic calcification | Calcification of muscle |
| Ectopic calcification | Calcinosis |
| Ectopic calcification | Calculus bladder |
| Ectopic calcification | Calculus prostatic |
| Ectopic calcification | Calculus ureteric |
| Ectopic calcification | Calculus urethral |
| Ectopic calcification | Calculus urinary |
| Ectopic calcification | Cardiac valve sclerosis |
| Ectopic calcification | Cerebral calcification |
| Ectopic calcification | Chondrocalcinosis |
| Ectopic calcification | Chondrocalcinosis pyrophosphate |
| Ectopic calcification | Cutaneous calcification |
| Ectopic calcification | Dystrophic calcification |
| Ectopic calcification | Heart valve calcification |
| Ectopic calcification | Heart valve stenosis |
| Ectopic calcification | Hepatic calcification |
| Ectopic calcification | Intervertebral disc calcification |
| Ectopic calcification | Intestinal calcification |
| Ectopic calcification | Ligament calcification |
| Ectopic calcification | Lymph node calcification |
| Ectopic calcification | Mitral valve calcification |
| Ectopic calcification | Mitral valve sclerosis |
| Ectopic calcification | Myocardial calcification |



| Category | PT |
|-----------------------|-------------------------------|
| Ectopic calcification | Nephrocalcinosis |
| Ectopic calcification | Nephrolithiasis |
| Ectopic calcification | Ovarian calcification |
| Ectopic calcification | Pancreatic calcification |
| Ectopic calcification | Pericardial calcification |
| Ectopic calcification | Pleural calcification |
| Ectopic calcification | Prostatic calcification |
| Ectopic calcification | Pulmonary calcification |
| Ectopic calcification | Pulmonary valve calcification |
| Ectopic calcification | Pulmonary valve sclerosis |
| Ectopic calcification | Splenic calcification |
| Ectopic calcification | Stag horn calculus |
| Ectopic calcification | Tendon calcification |
| Ectopic calcification | Tracheal calcification |
| Ectopic calcification | Tricuspid valve calcification |
| Ectopic calcification | Tricuspid valve sclerosis |
| Ectopic calcification | Vascular calcification |

# Restless legs syndrome:

| Category | PT |
|------------------------|---------------------------|
| Restless legs syndrome | Restless legs syndrome |
| Restless legs syndrome | Restlessness |
| Restless legs syndrome | Akathisia |
| Restless legs syndrome | Psychomotor hyperactivity |
| Restless legs syndrome | Sensory disturbance |
| Restless legs syndrome | Muscle cramp |
| Restless legs syndrome | Limb discomfort |
| Restless legs syndrome | Neuromuscular pain |
| Restless legs syndrome | Formication |



# **Appendix 5: Schedule of Events**

#### **Screening and Baseline Visits**

| | Screening <sup>1</sup> | | | | Baseline | 21 |
|---|---|---|---|---|---|---|
| VISIT TYPE/NUMBER | | TC 1 | TC 2 | | V1 | |
| STUDY WEEK or DAY | Week -4 | Week -3 | Week -1 | Day -2 | Day -1 | Day/Wk 0 |
| Informed Consent, Inclusion/Exclusion Criteria | X | | | | | |
| Medical History, Demographics, Height <sup>2</sup> | X | | | | | |
| PHEX Mutation Analysis 3,4 | | | | X | | |
| Tetracycline HCl or Demeclocycline Label <sup>5</sup> | | X | X | | | |
| Bone Biopsy <sup>1</sup> | | | | | X | |
| Bone Turnover Markers <sup>6</sup> | | | | X | | |
| Serum Phosphorus, Calcium, iPTH, Creatinine/eGFR <sup>6</sup> | X | | | X | | |
| Serum 1,25(OH) <sub>2</sub> D <sup>6</sup> | | | | X | | |
| Serum iFGF23 | $X^4$ | | | X | | |
| 2-hr Urine <sup>6,7</sup> | X | | | X | | |
| 24-hr Urine <sup>6,7</sup> | | | | X | | |
| BPI, BFI <sup>8,9</sup> | X | | | X | | |
| Skeletal survey <sup>10</sup> | | | | X | | |
| Anti-KRN23 (HAHA) | | | | | | X |
| Vital Signs 11 | X | | | X | X | X |
| Physical Examination | X | | | X | | |
| Weight <sup>12</sup> | | | | X | | |
| Renal Ultrasound <sup>1</sup> | X | | | | | |
| ECHO, ECG <sup>1</sup> | | | | X | | |
| Chemistry, Hematology (with PT/PTT), Urinalysis/pregnancy test <sup>6, 13, 14</sup> | X | | | X | | |
| Concomitant Medications | X | | | X | X | X |
| Adverse Events | X | | | X | X | X |
| KRN23 Administration | | | | | | X |




# **Open Label Treatment Period (Weeks 1 – 48)**

| VISIT TYPE/NUMBER <sup>15</sup> | HH<br>V2 | V3 | V4 | HH<br>V5 | HH<br>V6 | V7 | HH<br>V8 | HH<br>V9 | HH<br>V10 | HH<br>V11 | V12 | V13 | HH<br>V14 | HH<br>V15 | V16 | HH<br>V17 | HH<br>V18 | TC<br>3 | TC<br>4 | V1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WEEK | 1 | 2 | 4 | 6 | 8 | 12 | 14 | 16 | 20 | 21 | 22 | 24 | 28 | 32 | 36 | 40 | 44 | 45 | 47 | Day<br>1 | Day 2 |
| Tetracycline HCl or<br>Demeclocycline Label <sup>5</sup> | | | | | | | | | | | | | | | | | | X | X | | _ |
| Bone Biopsy <sup>1</sup> | | | | | | | | | | | | | | | | | | | | | $X^{16}$ |
| Bone Turnover Markers <sup>6</sup> | | | | | | X | | | | | | X | | | | | | | | X | |
| Serum Phosphorus, Calcium <sup>6</sup> | X | X | X | X | | X | X | | X | X | X | X | X | | X | | | | | X | |
| Serum 1,25(OH) <sub>2</sub> D <sup>6</sup> | X | X | X | | | | | | X | X | X | X | | | | | | | | X | |
| iPTH <sup>6</sup> | X | X | X | | | | | | X | X | X | | | | | | | | | X | |
| Serum iFGF23 <sup>6</sup> | | | | | | | | | | | | X | | | | | | | | X | |
| Serum Creatinine/eGFR <sup>6</sup> | | X | X | | | X | | | | | X | X | | | | | | | | X | |
| 2-hr Urine <sup>6,7</sup> | | X | X | | | X | | | | | X | X | | | | | | | | X | |
| 24-hr Urine <sup>6,7</sup> | | | | | | X | | | | | | X | | | X | | | | | X | |
| BPI, BFI 8,9 | | | | | | X | | | | | | X | | | X | | | | | X | |
| Targeted Radiography 10 | | | | | | X | | | | | | X | | | X | | | | | X | |
| KRN23 PK | X | X | X | | | | | | | X | X | X | | | | | | | | X | |
| Anti-KRN23 (HAHA) | | | X | | | | | | | | | X | | | | | | | | X | |
| Vital Signs 11 | | | X | | | X | | | | | | X | | | X | | | | | X | |
| Weight <sup>12</sup> | | | | | | X | | | | | | X | | | X | | | | | X | |
| Physical Examination | | | | | | X | | | | | | X | | | X | | | | | X | |
| Renal Ultrasound | | | | | | | | | | | | X | | | | | | | | X | |
| ECHO, ECG | | | | | | | | | | | | X | | | | | | | | X | |
| Chemistry, Hematology (with PT/PTT), Urinalysis <sup>6, 13</sup> | | | X | | | X | | | | | | X | | | X | | | | | X | |
| Urine Pregnancy Test 14 | | | X | | X | X | | X | X | | | X | X | X | X | X | X | | | X | |




| VISIT TYPE/NUMBER <sup>15</sup> | HH<br>V2 | V3 | V4 | HH<br>V5 | HH<br>V6 | V7 | HH<br>V8 | HH<br>V9 | НН<br>V10 | HH<br>V11 | V12 | V13 | HH<br>V14 | HH<br>V15 | V16 | НН<br>V17 | HH<br>V18 | TC<br>3 | TC<br>4 | V1 | 9 <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | | | | | | | 48 | ş <sup>1</sup> |
| WEEK | 1 | 2 | 4 | 6 | 8 | 12 | 14 | 16 | 20 | 21 | 22 | 24 | 28 | 32 | 36 | 40 | 44 | 45 | 47 | Day<br>1 | Day<br>2 |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | X | X |
| KRN23 ADMINISTRATION | | | X | | X | X | | X | X | | | X | X | X | X | X | X | | | X | |




## Treatment Extension Period (Weeks 49-96), Early Termination, and Safety Follow-up

| | Treatment Extension Period | | | | | | | | | | | | | | | Early Termination | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISIT TYPE/NUMBER <sup>15</sup> | HH<br>V20 | HH<br>V21 | V22 | HH<br>V23 | HH<br>V24 | HH<br>V25 | V26 | HH<br>V27 | HH<br>V28 | V29 | HH<br>V30 | HH<br>V31 | HH<br>V32 | V33 <sup>1</sup> | | ET <sup>1</sup> | Follow-up<br>Phone Call <sup>18</sup> | | |
| | | | | | | | | | | | | | | | TC 5 | | | 12 weeks | |
| WEEK | 52 | 56 | 60 | 64 | 68 | 70 | 72 | 76 | 80 | 84 | 88 | 92 | 94 | 96 | Week<br>-3 | Week<br>-1 | Day<br>1 | Day<br>2 | after Final<br>Dose <sup>18</sup> |
| Bone Biopsy <sup>1</sup> | | | | | | | | | | | | | | | | | | $X^{16}$ | |
| Tetracycline HCl or<br>Demeclocycline Label <sup>5, 16</sup> | | | | | | | | | | | | | | | X | X | | | |
| Bone Turnover Markers <sup>6</sup> | | | | | | | X | | | | | | | X | | | X | | |
| Serum Phosphorus, Calcium <sup>6</sup> | | | X | | | X | X | | | X | | | X | X | | | X | | |
| Serum 1,25(OH) <sub>2</sub> D <sup>6</sup> | | | X | | | X | X | | | X | | | X | X | | | X | | |
| iPTH <sup>6</sup> | | | X | | | X | X | | | X | | | X | X | | | X | | |
| Serum iFGF23 <sup>6</sup> | | | | | | | | | | | | | | X | | | X | | |
| Serum Creatinine/eGFR <sup>6</sup> | | | X | | | | X | | | X | | | | X | | | X | | |
| 2-hr Urine <sup>6,7</sup> | | | X | | | | X | | | X | | | | X | | | X | | |
| 24-hr Urine <sup>6,7</sup> | | | | | | | X | | | | | | | X | | | X | | |
| BPI, BFI <sup>8,9</sup> | | | | | | | X | | | | | | | X | | | | | |
| Targeted Radiography 10 | | | | | • | Only a | t clinic | visits | follow | ing a no | ewly di | iagnose | ed fract | ture <sup>17</sup> | | | | • | |
| Anti-KRN23 (HAHA) | | | | | | | X | | | | | | | X | | | X | | |
| KRN23 PK | | | | | | X | X | | | | | | | X | | | X | | |
| Vital Signs 11 | | | X | | | | X | | | X | | | | X | | | X | | |
| Weight <sup>12</sup> | | | | | | | X | | | | | | | X | | | X | | |
| Physical Examination | | | | | | | X | | | | | | | X | | | X | | |
| Renal Ultrasound | | | | | | | X | | | | | | | X | | | X | | |
| ECHO, ECG | | | | | | | X | | | | | | | X | | | $X^{17}$ | | |
| Chemistry, Hematology (with PT/PTT), Urinalysis <sup>6, 13</sup> | | | X | | | | X | | | X | | | | X | | | $X^{13}$ | | |
| Urine Pregnancy Test 14 | X | X | X | X | X | | X | X | X | X | X | X | | X | | | X | | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | X | X | X |


Study Number: UX023-CL304

Statistical Analysis Plan 15DEC 2016, Version 1.0



| | Treatment Extension Period | | | | | | | | | | | | | | | rly Tern | on | Safety<br>Follow-<br>up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISIT TYPE/NUMBER <sup>15</sup> | НН | НН | | НН | НН | НН | | НН | НН | | НН | НН | НН | | | Follow-up | | | |
| | V20 | V21 | V22 | V23 | V24 | V25 | V26 | V27 | V28 | V29 | V30 | V31 | V32 | V33 <sup>1</sup> | ET <sup>1</sup> | | | | Phone Call <sup>18</sup> |
| | | | | | | | | | | | | | | | TC 5 | TC 5 TC 6 ET | | | 12 weeks |
| WEEK | 52 | 56 | 60 | 64 | 68 | 70 | 72 | 76 | 80 | 84 | 88 | 92 | 94 | 96 | Week | Week | Day | Day | after Final |
| | | | | | | | | | | | | | | | -3 | -1 | 1 | 2 | Dose <sup>18</sup> |
| KRN23 | X | X | X | X | X | | X | X | X | X | X | X | | | | | | | |
| ADMINISTRATION | | | | | | | | | | | | | | | | | | | |

#### Footnotes to Table 2.1, Table 2.2, and Table 2.3

- The Baseline visit should occur no more than 31 days following the Screening visit. The bone biopsy must be completed on a day with no other procedures, and prior to dosing on Day 0. Renal ultrasound, ECHO, ECG, and x-rays may be performed within 3 days of indicated clinic visit to accommodate scheduling availability. The Baseline, Week 48, and Week 96 (or Early Termination; ET) assessments may be completed in any reasonable order (except where indicated) to allow for flexibility in scheduling. However, all Screening/Baseline assessments and inclusion/exclusion criteria must be satisfied prior to dosing.
- Medical history will include any available previous *PHEX* mutation analysis results for the subject or relevant family members with appropriate X-linked inheritance pattern. Height (in meters) will be obtained using a stadiometer (without shoes).
- <sup>3</sup> PHEX mutation analysis will be performed for all qualified subjects. If the Baseline result for PHEX mutation analysis is negative or inconclusive (i.e., No Mutation, Likely Benign, Variant of Uncertain Significance, or Possibly Pathogenic), and informed consent is provided by the subject, reflexive genetic testing will be performed to assess additional genes associated with phenotypes overlapping with XLH. A new blood sample for genetic analysis may be collected if necessary.
- For patients without prior *PHEX* mutation analysis who fail screening on the basis of the Kainos iFGF23 assay, *PHEX* analysis may be conducted before the baseline visit
- Available test results related to eligibility will be communicated to the subject within 1 week of the Screening visit by telephone call (TC1). If eligible, tetracycline HCl (or demeclocycline) will be provided to the subject with instructions for administration. The bone biopsy should be performed 5 days after the last dosing day for tetracycline or demeclocycline: The first dose should be given on days -20, -19, and -18 following TC1, and the second dose given on days -8, -7, and -6 following a second telephone call (TC2). The same instructions apply to TC3 and TC4 prior to the Week 48 (or TC5 and TC6 prior to ET if applicable) bone biopsy.
- Blood and urine to be collected after a minimum overnight fasting time of 8 hours and prior to drug administration (if applicable).
- Both 2-hr and 24-hr urine will be used for measurements of urinary phosphorus, creatinine and calcium; 2-hr urine will be used for the derivation of TmP/GFR and TRP.
- Only the BPI Question 3 (Worst Pain) will be administered at Screening for eligibility. The complete short-form BPI and BFI will be administered at all other indicated visits.
- Administer BPI first followed by BFI. The BPI and BFI should be administered prior to the performance of any invasive procedures.
- X-rays will be taken at locations pre-determined by skeletal survey (chest, lateral spine, right and left hand/wrist, right and left humerus, right and left radius/ulna, right and left femur/pelvis, right and left tibia/fibula, and right and left foot). If active pseudofracture(s) detected at baseline, targeted X-rays at

Study Number: UX023-CL304

Statistical Analysis Plan 15DEC 2016, Version 1.0



that location will be obtained as indicated. During the Extension Period, targeted x-rays will only be performed at clinic visit(s) to follow healing of any newly diagnosed fractures.

- Vital sign measurements consist of seated systolic/diastolic BP measured in millimeters of mercury (mm Hg; 2 measurements separated by 15 minutes), HR (beats per minute), respiration rate (breaths per minute), and temperature in degrees Celsius (°C). Obtain at the beginning of the visit before any additional assessments are completed
- Weight will be recorded in kilograms. Dose of study drug must be adjusted if weight increases by more than 20% from baseline.
- Serum chemistry panels may include PD parameters (i.e. serum phosphorus), and safety parameters of interest (i.e. calcium) to avoid duplication of testing. Screening and Week 48 Day1 hematology will include Prothrombin time/Partial thromboplastin time (PT/PTT). ET hematology will include PT/PTT if a bone biopsy is also scheduled (if a subject discontinues the study between 24 and 48 weeks)
- Urine pregnancy test for women of childbearing potential only. A serum pregnancy test will be performed in the event of a positive or equivocal urine pregnancy test result.
- During the Open-Label Treatment Period (Weeks 1 48) and Treatment Extension Period (Weeks 49-96) subjects will return to the clinic and/or have home health (HH) visits as indicated (± 5 days). HH visits may also be conducted at the clinic depending on subject proximity to the investigational site and local availability of home health care resources.
- Bone biopsies will not be performed at Week 48 (or at ET) for subjects who do not have evidence of osteomalacia on the initial biopsy. Bone biopsies will not be performed at the ET Visit if the subject discontinues within 6 months of the baseline biopsy or if the subject terminates the study after 48 weeks. Prior to ET biopsy, tetracycline HCl (or demeclocycline) will be provided to the subject with instructions for administration. The bone biopsy should be performed 5 days after the last dosing day for tetracycline or demeclocycline The first dose should be given on days -20, -19, and -18 following TC5, and the second dose given on days -8, -7, and -6 following a second telephone call (TC6) prior to the ET biopsy (if eligible).
- Targeted X-rays and ECHO will not be performed at ET if the assessment was conducted within 3 months of termination. Targeted X-rays will not be taken at ET if the subject terminates the study after 48 weeks.
- To be completed only for subjects who complete the study and choose not to enroll in a planned extension study under a separate protocol or subjects who discontinue the study early. This call is not required for subjects who are eligible and choose to participate in the separate extension study. The site personnel will initiate this safety follow-up telephone call 12 weeks ± 5 days after a subject's last dose of study drug to collect information on any ongoing or new AEs, serious adverse events (SAEs), and concomitant medications. Appropriate follow-up should continue until all safety concerns, in the Investigator's opinion, are resolved.